CLINICAL TRIAL: NCT02658591
Title: Effects of Faba Bean Fractions as Ingredients in Novel Food Products on Glycemia, Appetite and Metabolic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SPG_UofT_FabaBean
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Diabetes
Keywords: Food intake; Satiety; Appetite; Glycemia; Faba bean; Protein; Snack
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (Active Comparator): Crackers/pasta with no faba bean fraction
  Interventions: Dietary Supplement: Crackers/pasta with no faba bean fraction
- Faba bean protein concentrate (Experimental): Crackers/pasta with added faba bean protein concentrate
  Interventions: Dietary Supplement: Crackers/pasta with added faba bean protein concentrate
- Faba bean protein isolate (Experimental): Crackers/pasta with added faba bean protein isolate
  Interventions: Dietary Supplement: Crackers/pasta with added faba bean protein isolate
- Faba bean flour (Experimental): Crackers/pasta with added faba bean flour
  Interventions: Dietary Supplement: Crackers/pasta with added faba bean flour
- Faba bean starch (Experimental): Crackers/pasta with added faba bean starch
  Interventions: Dietary Supplement: Crackers/pasta with added faba bean starch

INTERVENTIONS:
Dietary Supplement: Crackers/pasta with added faba bean protein concentrate — Protein concentrate treatment
  Arms: Faba bean protein concentrate
Dietary Supplement: Crackers/pasta with added faba bean protein isolate — Protein isolate treatment
  Arms: Faba bean protein isolate
Dietary Supplement: Crackers/pasta with added faba bean starch — Starch treatment
  Arms: Faba bean starch
Dietary Supplement: Crackers/pasta with added faba bean flour — Flour treatment
  Arms: Faba bean flour
Dietary Supplement: Crackers/pasta with no faba bean fraction — Control treatment
  Arms: Control

SUMMARY:
The investigators hypothesized that consuming crackers or pasta enriched with faba bean fractions (faba bean protein concentrate, faba bean protein isolate, faba bean flour and faba bean starch), would reduce the blood glucose response to the meal compared to foods without faba bean components and reduce food intake at a meal

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* No metabolic disease
* BMI 20 - 25 kg/m^2
* Male
* Age 18-30

Exclusion Criteria:

* Intolerance to treatments
* Currently taking appetite-modifying medications
* Restrictive eating
* Smoking
* Over- or underweight
* Breakfast-skipping

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose levels | Starting at the beginning of each session (0 minutes, before consumption of treatment) and every 15 - 30 minutes up to 200 minutes (time of completion of each session)
  Each participant will attend 5 sessions in total (randomized 5-arm cross-over design)
Change in gut hormone levels measured in the blood | Starting at the beginning of each session (0 minutes, before consumption of treatment) and every 30 minutes up to 200 minutes (time of completion of each session)
  Each participant will attend 5 sessions in total (randomized 5-arm cross-over design)

SECONDARY OUTCOMES:
Subjective appetite | From 0 to 200 minutes
  Measured using Visual Analog Scales (VAS)
Ad libitum food (pizza meal) intake as measured by the amount of pizza (in grams) consumed during the 20 minute period | 120 minutes after completion of treatment, 20 minutes were allocated to allow for pizza consumption
  Each participant will also answer questions related to physical comfort, motivation to eat, and rating feelings of energy and fatigue using Visual Analog Scales (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chan CKY, Fabek H, Mollard RC, Jones PJH, Tulbek MC, Chibbar RN, Gangola MP, Ramadoss BR, Sanchez-Hernandez D, Anderson GH. Faba bean protein flours added to pasta reduce post-ingestion glycaemia, and increase satiety, protein content and quality. Food Funct. 2019 Nov 1;10(11):7476-7488. doi: 10.1039/c9fo01186b. Epub 2019 Oct 31. PMID 31670336